CLINICAL TRIAL: NCT03176563
Title: Observational Study of Patients With Uncomplicated Urinary Tract Infection Treated With Antibiotics or Herbal Medicinal Product
Brief Title: Observational Follow-up Study of REGATTA
Acronym: REGATTA II
Status: Completed | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Karsten Gavenis, Quality Assurance Staff Unit Clinical Trials, University Medical Center Goettingen
Other Study IDs: 01970
Record Dates: First submitted 2017-05-31; First posted 2017-06-05 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Urinary Tract Infections
Keywords: herbal treatment; antibiotics; uncomplicated urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Fosfomycin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women treated with the herbal drug Uva Ursi: Patients of the clinical trial REGATTA (NCT03151603) who have been randomized in the Uva Ursi arm.
  Interventions: Drug: Arctuvan; Drug: Placebo to Fosfomycin
- Women treated with antibiotics: Patients of the clinical trial REGATTA (NCT03151603) who have been randomized in the fosfomycin arm.
  Interventions: Drug: Fosfomycin; Drug: Placebo to Arctuvan

INTERVENTIONS:
Drug: Arctuvan — application of a herbal drug in the clinical trial REGATTA (NCT03151603)
  Groups: Women treated with the herbal drug Uva Ursi
Drug: Placebo to Fosfomycin — application of Placebo to Fosfomycin in the clinical trial REGATTA (NCT03151603)
  Groups: Women treated with the herbal drug Uva Ursi
Drug: Fosfomycin — application of an antibiotic drug in the clinical trial REGATTA (NCT03151603)
  Groups: Women treated with antibiotics
Drug: Placebo to Arctuvan — application of Placebo to Arctuvan in the clinical trial REGATTA (NCT03151603)
  Groups: Women treated with antibiotics

SUMMARY:
Observational follow-up study of patients included in the clinical trial REGATTA.

DETAILED DESCRIPTION:
A follow-up telephone interview of the participants of the clinical trial REGATTA exploring the occurrence of urinary tract infections, pyelonephritis within a follow-up period of three months after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* participants of the clinical trial REGATTA
* informed consent to participate in the observational study REGATTA II

Exclusion Criteria:

- no informed consent granted

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: participants of the clinical trial REGATTA
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
number of urinary tract infections | 3 months after inclusion in REGATTA
  number of urinary tract infection within 3 months after inclusion in REGATTA
number of pyelonephritis | 3 months after inclusion in REGATTA
  number of pyelonephritis within 3 months after inclusion in REGATTA

CONTACTS AND LOCATIONS:
Overall Officials: Eva Hummers-Pradier, Prof. Dr., Principal Investigator — University Medical Center Göttingen
Locations (47):
- Germany (47):
  - Hausarztpraxis Dr. Raby, Achim
  - General Practice Aden, Braunschweig
  - General Practice Scheffer, Braunschweig
  - General Practice Coutelle, Bremen
  - General Practice Schelp, Bremen
  - General Practice Dickow, Burgwedel
  - General Practice Kiwit-Putzer, Burgwedel
  - Praxis Zietz, Celle
  - General Practice Kutzsche, Emmerthal
  - Praxis Dr. Bahr, Gieboldehausen
  - General Practice Müller, Gillersheim
  - Institute of General Medicine, University Medical Center Goettingen, Goettigen
  - General Practice Keske, Göttingen
  - General Practice Koch, Göttingen
  - General Practice Kolb, Göttingen
  - General Practice Lang, Göttingen
  - General Practice Lückerath, Göttingen
  - Praxisgemeinschaft Jacob / Kling, Göttingen
  - Institute of General Medicine, MHH Hannover, Hanover
  - General Practice Barth, Hanover
  - Praxis Dr. Egner, Hanover
  - General Practice Löber, Hardegsen
  - Gemeinschaftspraxis Dres Schlesier / Eckhardt, Heilbad Heiligenstadt
  - Gemeinschaftspraxis Hartleb / Stöcking, Heilbad Heiligenstadt
  - Praxis Dr. Koch, Heilbad Heiligenstadt
  - Praxisgemeinschaft Seitz / Eckert, Herzberg am Harz
  - General Practice Wilde, Hildesheim
  - General Practice Beverungen, Höxter
  - Praxisgemeinschaft Stoltz / Raddatz, Höxter
  - Gemeinschaftspraxis Kasperczyk / Schindewolf-Lensch, Isernhagen-Süd
  - General Practice Franz, Katlenburg-Lindau
  - Praxis Dr. Ohlendorf, Langenhagen
  - General Practice Ertel, Langwedel
  - General Practice Wehrbein, Lemförde
  - General Practice Lindenblatt, Neustadt
  - Hausarztzentrum Nörten, Nörten-Hardenberg
  - General Practice Preiskorn, Rehburg-Loccum
  - General Practice Meier-Ahrens, Rosdorf
  - General Practice Woitschek, Salzgitter
  - General Practice Beulshausen, Sattenhausen
  - General Practice Schulte, Scheeßel
  - General Practice Böttcher, Schwanewede
  - General Practice Albrecht, Springe
  - General Practice Wolf, Uslar
  - General Practice Schmiemann, Verden an der Aller
  - General Practice Annweiler, Waake
  - General Practice Stegemann, Wunstorf